CLINICAL TRIAL: NCT06129981
Title: Treatment of Post-traumatic Stress Disorder by Exposure Psychotherapy in Augmented Imagination by Vocal Feedback : Acceptability Study
Brief Title: TREATMENT OF POST-TRAUMATIC STRESS DISORDER USING AUGMENTED IMAGINATION EXPOSURE PSYCHOTHERAPY WITH VOCAL FEEDBACK: AN ACCEPTABILITY STUDY
Acronym: TRAUMAVOICE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022_0525; 2022-A02423-40 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2023-08-21; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-01

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Post-traumatic stress disorder; Augmented Therapy; Voice Transformations; Algorithms
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaginary exposure therapy augmented by vocal feedback in patients fulfilling the criteria for PTSD (Experimental)
  Interventions: Behavioral: Imaginary exposure therapy augmented by vocal feedback

INTERVENTIONS:
Behavioral: Imaginary exposure therapy augmented by vocal feedback — The procedure specific to the study
  * adding inclusion procedures (explanation of the study, verification of inclusion and non-inclusion criteria, signature of informed consent)
  * including, in the usual initial V0 visit, psychometric measures specific to the study (RSDI, CGI, PMI, GEW)
  * including a single usual psychotherapy session (i.e. not augmented) S1, during which the psychometric (RSDI, PMI, GEW) and psychophysiological (connected watch) measurements specific to the study are used
  * adding the VF device and using psychometric (RSDI, PMI, GEW) and psychophysiological (connected watch) measurements specific to the study during psychotherapy sessions S2 to Sn (minimum S6)
  * adding, during the last usual end-of-treatment visit, psychometric measures specific to the study (CGI)
  * adding psychometric measures specific to the study during the usual follow-up visit at 3 months
  * adding a follow-up visit at 12 months (CGI, PCL-5), either by telephone or on-site.

SUMMARY:
We now have many pharmacological and psychotherapeutic treatments for patients suffering from Post Traumatic Stress Disorder (PTSD), including cognitive and behavioral therapy (CBT) by reactivation of traumatic memories. Despite remarkable initial efficacy, only one-third of patients treated with CBT show lasting clinical improvement. On the other hand, the associated drop-out rates vary from 17% to 33%, which may be linked to the difficulty of the task, which implies reactivating the traumatic memory (Bradley et al. 2005).

Alternative treatments for PTSD include blocking chemo-facilitated memory reconsolidation with a beta-blocker, propranolol. Briefly, reconsolidation theory posits that a recalled memory becomes unstable again before consolidating again into long-term memory, hence the term "reconsolidation". During this phase of transitory plasticity, the memory can be modulated, in particular its emotional charge. The use of propranolol has shown its benefit during this phase in patients suffering from PTSD (Brunet et al, 2018). However, the use of this facilitated chemo therapy is limited to patients with no contraindication to taking beta-blockers. In this context, a non-medicinal alternative to attenuate the emotional strength of the memory has a therapeutic interest.

One of the ways in which our emotional experience can be modulated is through the perception of our emotional behavior. According to the theory of self-perception (Bem, 1972) individuals become aware or conscious of their attitudes, emotions and other internal states in part by inferring them from the observation of their own behaviors. Thus when individuals produce sounds or facial expressions typical of specific emotions such as joy, sadness or anger, they will tend to experience an emotional state congruent with their vocal or facial production (Hatﬁeld and Hsee, 1995).

Work on the influence of voice perception, in particular, is experiencing a new boom due to technical developments in the fields of acoustic signal processing. In particular, Dr. Aucouturier's team has created a software device to directly modify the emotional tone of speech formulated orally. For example, for "happy" manipulation, the pitch of the voice is changed with a pitch shifting algorithm to make it more positive, the dynamic range of the voice is increased with a compression algorithm to make it more confident, and its spectral content is modified with a high-pass filter to make it brighter. The results of this work (Aucouturier et al. 2016; Rachman et al. 2018; Goupil et al., 2021) showed an emotional vocal feedback effect: the subjective evaluation that participants make of their emotional state after modification by the device goes in the direction of the emotion created by the platform, even though the participants are typically unaware of the operated modulation. The non-detection of the transformation being a necessary condition for observing the effect of VF on the emotional state of the participant.

The rationale of this study is to test the use of a real-time vocal transformation paradigm during exposure therapy by reactivation of traumatic memory in imagination in patients. During this therapy, the patient is asked to read aloud the very detailed script of the traumatic event. We want to test whether manipulating the emotional tone of the patient's voice online, when reading, can have a facilitating impact on the process of reducing the emotional charge associated with the traumatic script. In order to justify the use of the audio headphones as well as the microphone, and to ensure us of the non-detectability of the transformation operated on the voice, we will explain to our patients that this device (hearing his voice in a headphone during the session of re-exposure to a memory) aims to increase immersion. Our main objective will be to assess the acceptability of this augmented form of psychotherapy, and our secondary objectives will be to assess its technical feasibility and provide initial elements to assess its effectiveness. The results will be compared with data from the literature on the usual treatment (imaginary exposure therapy, with or without propranolol according to the indications).

ELIGIBILITY:
Inclusion Criteria:

* Male or female over the age of 18
* Meeting DSM-5 criteria for Post-Traumatic Stress Disorder
* Presenting a PCL-5 strictly greater than 32 (PCL-5, Weathers et al., 2013)
* Giving consent by signing the consent form after clear and honest information about the study.
* Being able to understand, speak and read French

Exclusion Criteria:

* Deaf, dumb or hearing aid patient
* Minors or adults under guardianship or curatorship, under judicial protection, persons deprived of liberty
* Suffering from a bipolar or psychotic disorder
* Having suffered a head trauma for less than a year or having clinical symptoms and carrying neurological sequelae
* Presenting a proven severe suicidal risk (Mini-International Neuropsychiatric Interview-Suicidality module, MINI-S and medical examination)
* Suffering from a substance use disorder (MINI-DSM5)
* Being treated for less than 2 months with antidepressants
* Not being affiliated to a social security scheme
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
assess whether the use of the vocal feedback (VF) device during imaginative exposure psychotherapy is acceptable for patients with PTSD. | For the duration of the study for each patient; i.e. 12 months
  Patient compliance with VF-enhanced exposure psychotherapy evaluated by the drop-out rate, including loss of sight of patients who do not show up for the scheduled session and no longer respond to the solicitations of the clinical team, and the discontinuation of patients who express the wish to withdraw from the study.

SECONDARY OUTCOMES:
Assess other aspects of the acceptability of the VF system: assess the evolution of patients' motivation | Throughout the duration of therapy for the patient + the initial V0 visit, i.e. an average of 7 weeks, or even a few weeks more depending on the number of sessions required to sufficiently reduce PTSD symptoms (PCL-5 < 33).
  The patient's motivation after each session is assessed by the Patient Motivation Inventory questionnaire (PMI; Gudjonsson et al., 2007)
Assess other aspects of the acceptability of the VF system: - evaluate the evolution of patients' emotional feelings | Throughout the duration of therapy for the patient + the initial V0 visit, i.e. an average of 7 weeks, or even a few weeks more depending on the number of sessions needed to sufficiently reduce PTSD symptoms (PCL-5 < 33).
  The patient's emotional feelings are assessed by the "effective re-experience" subscale of the Responses to Script-Driven Imagery Scale (RSDI) questionnaire (Hopper et al., 2007a).
Assess the feasibility of the VF system: assess the ability of the VF device to acoustically modify the patient's voice in the direction of an attenuation of the negative emotional tone | For the entire duration of VF-enhanced exposure therapy, i.e. an average of 5 weeks per patient, or even a few weeks more depending on the number of sessions required to sufficiently reduce PTSD symptoms (PCL-5 < 33)
  The ability of the VF device to acoustically alter the patient's voice in the direction of an attenuation of the negative emotional tone is assessed by making an audio recording of the patient's voice entering and exiting the device (i.e. before and after transformation), and by performing an automated acoustic analysis with the PRAAT software (https://www.fon.hum.uva.nl/praat/). The acoustic characteristics extracted are the pitch (average, standard deviation, minimum and maximum), jitter (quantifying the fluctuations of the fundamental period of the signal from one cycle to another: local, absolute, relative average disturbance, period disturbance quotient) and the shimmer (local amplitude variations) between two consecutive periods (local, localdB, over 3, 5 and 11 periods and the proportion of noise in the signal (Noise-to-harmonic ratio, Harmonic-to-noise ratio).
Assess the feasibility of the VF system: assess the rate of detectability by the patient of the vocal transformation applied to his voice during VF-enhanced psychotherapy | For the entire duration of VF-enhanced exposure therapy, i.e. an average of 5 weeks per patient, or even a few weeks more depending on the number of sessions needed to sufficiently reduce PTSD symptoms (PCL-5 < 33).
  Patients' detectability of the vocal transformation is assessed on the basis of a debriefing carried out by the caregiver at the end of each session with increasingly specific questions concerning the sound quality and the voice heard by the patient: " what did you think of the device? / "How did you find the sound quality?" / "how did you find the sound of your voice?". Patients' answers to these open-ended questions are recorded and then scored after the session by the psychologist on a scoring grid ranging from 1 = "you intentionally transformed my voice during this session", 2: "my voice was sometimes higher or lower than usual during this session", 3: "my voice sounded strange during this session", 4: "my voice sounded strange, but it's probably because I don't have the used to hearing my voice through headphones", 6: "my voice was as usual". Scores 1-3 are considered transformation detection.
provide initial elements for evaluating the effectiveness of the device on the reduction of post-traumatic symptoms: assess the evolution of PTSD symptoms after S6 (or Sn, n being defined by the PCL-5<33 criterion) | Throughout the duration of the study for each patient, i.e. 12 months.
  The evolution of PTSD symptoms in patients receiving VF-augmented therapy is assessed with the PCL-5 questionnaire, self-administered pre-treatment, at the start of each S1-Sn session, then post-treatment (visit end of treatment, then follow-up visits at 3 and 12 months), the percentage of diagnosis of PTSD (PCL-5 questionnaire threshold > 32) pre- versus post-treatment, and the average number of sessions required to go below the score threshold.
Evaluating the effectiveness of the device on the reduction of post-traumatic symptoms: assess the relapse rate at 3 and 12 months (after W6 or Sn, n being defined by the PCL-5<33 criterion) of patients receiving VF-enhanced therapy | Measurement at 3 and 12 months for each patient.
  The relapse rate at 3 months and 12 months of patients receiving VF-augmented therapy is assessed by comprehensive clinical assessment including clinical global assessment (CGI) and PTSD symptom assessment (PCL-5)
Evaluating the effectiveness of the device on the reduction of post-traumatic symptoms: assess the evolution of patients' heart rate variability (HRV) during each VF-augmented therapy session (S1 to S6 or Sn), and from session to session | Throughout the duration of therapy for each patient, i.e. 6 weeks on average, or even a few weeks longer depending on the number of sessions required to sufficiently reduce PTSD symptoms (PCL-5 < 33).
  The evolution of patients' HRV during each VF-enhanced therapy session will be measured with an EMPATICA connected watch, worn on the patient's wrist during the session
Provide the first clustering elements of patients' characteristics according to their response to the device: assess the correlation of effectiveness measures and device feasibility measures | During the entire duration of therapy for the patient + the initial V0 visit, i.e. an average of 7 weeks, or even a few weeks more depending on the number of sessions needed to sufficiently reduce PTSD symptoms (PCL-5 < 33).
  Assess the correlation between efficacy criteria (symptoms, relapse, HRV) and the feasibility criteria (detection, acoustic intensity of the transformation)
provide initial clustering elements of patient characteristics according to their response to the device: assess the influence of dissociative symptoms on the feasibility and effectiveness of the device | measurements collected over the entire duration of the study for each patient, i.e. 12 months. However, a preliminary analysis can be made at the end of the therapy period, which will last an average of 7 weeks
  patients' dissociative symptoms at pre-treatment with the dissociation subscale of the Responses to Script-Driven Imagery Scale (RSDI) questionnaire (Hopper et al., 2007). These symptoms will be used for a differential analysis assessing their influence on the above-mentioned measures of effectiveness and feasibility.
Provide the first clustering elements of patients' characteristics according to their response to the device: - highlight the characteristics (severity of initial symptoms) of "responders" and "non-responders". | measurements collected over the entire duration of the study for each patient, i.e. 12 months. However, a preliminary analysis can be made at the end of the therapy period, which will last an average of 7 wekks
  To provide initial clustering elements of patient characteristics according to their response to the device, we will assess: the "responder" or "non-responder" status of patients with the following criterion: PCL<33 at S6, or >20-30% improvement in symptoms.